CLINICAL TRIAL: NCT03171805
Title: Post-balloon Occluded Retrograde Transvenous Obliteration Use of Propranolol for the Prevention of Worsening of Esophageal Varices in Patients With Isolated Gastric Varices
Brief Title: The Use of Propranolol for the Prevention of Worsening of Esophageal Varices in Patients With Isolated Gastric Varices
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, luo xuefeng, Attending doctor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Propranolol in GV
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Liver Cirrhoses; Portal Hypertension; Gastric Varix
MeSH Terms: conditions — Hypertension, Portal; Esophageal and Gastric Varices | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propranolol group (Experimental): Propranolol was given after patients with cirrhosis and isolated gastric varices underwent balloon occluded retrograde transvenous obliteration successfully.
  Interventions: Drug: Propranolol
- control group (No Intervention): Propranolol was not given after patients with cirrhosis and isolated gastric varices underwent balloon occluded retrograde transvenous obliteration successfully.

INTERVENTIONS:
Drug: Propranolol — Propranolol was given after patients with cirrhosis and isolated gastric varices underwent balloon occluded retrograde transvenous obliteration successfully.
  Arms: Propranolol group

SUMMARY:
Balloon-occluded retrograde transvenous obliteration (BRTO) has been effective method to manage gastric varices. However, more than one third of patients after BRTO treatment experienced worsening of esophageal varices. The present study was designed to evaluate the effect of post-BRTO propranolol adminstration on the change of esophageal varices.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of liver cirrhosis
2. Clinical diagnosis of isolated gastric varices
3. The presenec of spontaneous portosystemic shunt

Exclusion Criteria:

1. Contradictions to Propranolol
2. Balloon occluded retrograde transvenous obliteration was failed

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2022-05-15 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Worsening of esophageal varices rate | 3 years
  Analysis

SECONDARY OUTCOMES:
Variceal rebleeding rate | 3 years
  Analysis
Mortality rate | 3 years
  Analysis
Worsening of ascites rate | 3 years
  Analysis

CONTACTS AND LOCATIONS:
Overall Officials: xuefeng luo, Principal Investigator — Sichuan University
Locations (1):
- West china Hospital, Chengdu, China

IPD SHARING:
Plan to Share IPD: Undecided